CLINICAL TRIAL: NCT05601193
Title: Effect of Ovarian Injection of Autologous Platelet-Rich Plasma on the Pregnancy Outcome of IVF/ICSI in Patients With Poor Ovarian Response: A Prospective Randomized Controlled Study
Brief Title: Ovarian PRP Injection in Women With POR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022ZSLYEC-495
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Poor Ovarian Response
Keywords: Poor Ovarian Response; Platelet-Rich Plasma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): Experimental: autologous PRP Bilateral ovaries autologous PRP injection under transvaginal ultrasound guidance. 3ml on each ovary.Once a month. two consecutive injections
  Interventions: Other: autologous platelet-rich plasma
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: autologous platelet-rich plasma — autologous PRP preparation was done by segregation of PRP following the centrifugation
  Arms: PRP group

SUMMARY:
Patients with poor ovarian response (POR）is considered one of most challenging tasks in artificial reproductive treatment (ART). Several retrospective studies have shown that platelet-rich plasma (PRP) is one of the proposed therapeutic strategies for women with POR. However, prospective randomized controlled trials are still lacking. This study aimed to evaluate the effect on intraovarian injection of autologous PRP in poor ovarian reserve prospectively.

DETAILED DESCRIPTION:
It will be divided two groups of POR patients according to the treatment itself. One group was treated by intraovarian injection of autologous PRP, and the other was control. It will detect the function of ovarian reserve and IVF outcomes before and after treatment in both two groups. In addition, granulosa cells and follicular fluid before and after injection were collected for functional exploration experiments.

ELIGIBILITY:
Inclusion Criteria:

* 1) Women less than 43 years old and undergo IVF/ICSI; 2) AMH < 1.1 and the number of follicles in bilateral antrum < 7; 3) those who have obtained less than or equal to 3 follicles in conventional controlled ovulation cycle or whose diameter ≥ 14mm on the trigger day; or have a previous history of ovarian cyst removal; if the woman is less than 40 years old, she needs to meet the inclusion criteria 2 and 3 at the same time. If you are 40 years old or older, you can join the group if you meet the inclusion criteria 2 or 3.

Exclusion Criteria:

* 1) patients with clear indications or plans to undergo pre-embryo transfer genetic diagnosis (PGD) and preimplantation genetic screening (PGS); 2) patients with recurrent abortion who had more than 2 consecutive spontaneous abortions (including biochemical pregnancy); 3) men with azoospermia who underwent microsemen extraction; 4) benign ovarian cysts (endometriosis cyst, teratoma, etc.) found by B-ultrasound; 5) women with heart, liver and kidney insufficiency. 6) one of the husband and wife has chromosome abnormality; 7) the history of malignant tumor of the woman or the hereditary family history of the husband and wife 8) uterine anatomical abnormalities (including uterine adhesion, endometrial polyps, submucous myoma, uterine mediastinum, etc.) 9) untreated hydrosalpinx 10) uncontrolled endocrine abnormalities, including thyroid dysfunction, diabetes, etc. 11) other reasons that the researchers believe are not appropriate to participate in this study, such as positive for syphilis or HIV.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 390 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
number of oocytes retrieval | 2 years
  The number of oocytes retrieval under the same ovarian stimulation protocol before and after PRP injection

SECONDARY OUTCOMES:
Ovarian function in DOR patients before and after PRP injection. | 2 years
  Anti-müllerian Hormone (AMH) serum level, Follicle Stimulating Hormone (FSH) serum level, Estradiol (E2) serum level level on menstrual day 2/3
Outcomes of IVF in DOR patients before and after PRP injection under the same ovarian stimulation protocol. | 3 years
  The number of oocyte retrieval, fertilization rate , blastocyst formation rate, implantation rate, incidence of clinical pregnancy rate

OTHER OUTCOMES:
Functional experiments of follicular fluid and granulosa cells before and after PRP injection | 1 year
  Changes of hormone/ RNA/ protein / growth factor expression in follicular fluid and granulosa cells before and after PRP injection

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Research Center, the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China